CLINICAL TRIAL: NCT00620113
Title: A Randomized, Double-Blind, Placebo-Controlled, Parallel-Group, Multicenter Dose-Finding Study of MK-0822 in the Treatment of Involutional Osteoporosis
Brief Title: Efficacy and Safety of Odanacatib (MK-0822) in Participants With Involutional Osteoporosis (MK-0822-022)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0822-022; MK-0822-022 (Other: Merck Registration Number); 2007_034 (Other: Merck)
Record Dates: First submitted 2008-01-29; First posted 2008-02-21 (Estimated); Results first posted 2017-03-13 (Actual); Last update posted 2018-08-27 (Actual); Status verified 2018-07

CONDITIONS: Osteoporosis Postmenopausal
MeSH Terms: conditions — Osteoporosis, Postmenopausal | interventions — odanacatib; Cholecalciferol; Calcium Carbonate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Placebo (Placebo Comparator): After an observation period of ~5 weeks, participants receive dose-matched placebo to odanacatib once weekly for 52 weeks. Participants also receive weekly supplementation with open-label 5600 International Units (IU) vitamin D3 and 500 mg of open-label daily calcium supplement (if calcium <1000 mg per day from dietary and other sources) throughout the observation and treatment periods.
  Interventions: Dietary Supplement: Vitamin D3; Dietary Supplement: Calcium carbonate; Drug: Placebo
- Odanacatib 10 mg (Experimental): After an observation period of ~5 weeks, participants receive 10 mg odanacatib once weekly for 52 weeks. Participants also receive weekly supplementation with open-label 5600 IU vitamin D3 and 500 mg of open-label daily calcium supplement (if calcium <1000 mg per day from dietary and other sources) throughout the observation and treatment periods.
  Interventions: Drug: Odanacatib; Dietary Supplement: Vitamin D3; Dietary Supplement: Calcium carbonate
- Odanacatib 25 mg (Experimental): After an observation period of ~5 weeks, participants receive 25 mg odanacatib once weekly for 52 weeks. Participants also receive weekly supplementation with open-label 5600 IU vitamin D3 and 500 mg of open-label daily calcium supplement (if calcium <1000 mg per day from dietary and other sources) throughout the observation and treatment periods.
  Interventions: Drug: Odanacatib; Dietary Supplement: Vitamin D3; Dietary Supplement: Calcium carbonate
- Odanacatib 50 mg (Placebo Comparator): After an observation period of ~5 weeks, participants receive 50 mg odanacatib once weekly for 52 weeks. Participants also receive weekly supplementation with open-label 5600 IU vitamin D3 and 500 mg of open-label daily calcium supplement (if calcium <1000 mg per day from dietary and other sources) throughout the observation and treatment periods.
  Interventions: Drug: Odanacatib; Dietary Supplement: Vitamin D3; Dietary Supplement: Calcium carbonate

INTERVENTIONS:
Drug: Odanacatib — Odanacatib tablets 10 mg, 25 mg, or 50 mg (depending upon randomization), taken orally once weekly for 52 weeks.
  Other Names: MK-0822
  Arms: Odanacatib 10 mg; Odanacatib 25 mg; Odanacatib 50 mg
Dietary Supplement: Vitamin D3 — Two Vitamin D3 tablets (5600 IU total) taken orally once weekly for 52 weeks.
  Other Names: cholecalciferol
Dietary Supplement: Calcium carbonate — Calcium carbonate 500 mg tablet taken orally every day for 52 weeks.
Drug: Placebo — Dose-matched placebo tablets to odanacatib, taken orally once weekly for 52 weeks.
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess the dose-response on the percent change from baseline in lumbar spine bone mineral density (BMD) at lumbar vertebrae 1 to 4 (L1- L4) when odanacatib (MK-0822) 10 mg, 25 mg, 50 mg or placebo is orally administered once weekly for 52 weeks to Japanese involutional osteoporosis participants. The study will also assess safety and tolerability of odanacatib (10, 25, and 50 mg) in these participants.

The study will enroll approximately 280 participants and randomly assign them to 3 different doses of odanacatib or placebo for 52 weeks, along with supplemental vitamin D3 and calcium carbonate. The primary efficacy hypothesis is that a dose-response relationship on the percent change from baseline in lumbar spine BMD (L1- L4) is seen when odanacatib 10, 25, 50 mg or placebo is orally administered once weekly for 52 weeks to involutional osteoporosis participants. The primary safety hypothesis is that odanacatib will be safe and well tolerated over 52 weeks to involutional osteoporosis participants.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal woman (for at least 5 years) or men who are aged between 45 to 85
* Participant who has low bone mineral density
* Participant has anatomy suitable for dual-energy x-ray absorptiometry (DXA) of the lumber spine and hip
* Participant is ambulatory (can walk)

Exclusion Criteria:

* Participant has secondary osteoporosis or has a metabolic bone disorder other than osteoporosis or osteopenia
* Participant has received osteoporosis medications or other medications that affect bone
* Participant is already participating in another drug study

Ages: 45 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 287 (Actual)
Dates: Start 2007-12-03 (Actual); Primary Completion 2009-05-29 (Actual); Study Completion 2009-05-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
https://www.merck.com/clinical-trials/pdf/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Background] Nakamura T, Shiraki M, Fukunaga M, Tomomitsu T, Santora AC, Tsai R, Fujimoto G, Nakagomi M, Tsubouchi H, Rosenberg E, Uchida S. Effect of the cathepsin K inhibitor odanacatib administered once weekly on bone mineral density in Japanese patients with osteoporosis--a double-blind, randomized, dose-finding study. Osteoporos Int. 2014 Jan;25(1):367-76. doi: 10.1007/s00198-013-2398-2. Epub 2013 May 29. PMID 23716037

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of 403 participants screened, 287 participants were randomized to treatment on study. 286 participants received the correct treatment on study and were used for safety and efficacy analyses. One participant in the odanacatib 25 mg group also received 50 mg odanacatib during study by mistake and was excluded from all analyses.
Period: Overall Study
Arm/Group | Placebo | Odanacatib 10 mg | Odanacatib 25 mg | Odanacatib 50 mg
Started | 73 | 74 | 71 (Includes 1 participant who also received 50 mg dose by accident during study.) | 69
Efficacy/Safety Population | 73 | 74 | 70 | 69
Completed | 60 | 67 | 66 (Includes 1 participant who also received 50 mg dose by accident during study.) | 59
Not Completed | 13 | 7 | 5 | 10
Not completed — Adverse Event | 3 | 2 | 2 | 1
Not completed — Lack of Efficacy | 2 | 3 | 0 | 2
Not completed — Physician Decision | 1 | 0 | 0 | 2
Not completed — Protocol Violation | 2 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 5 | 1 | 3 | 5

BASELINE CHARACTERISTICS:
Population: Safety Population: All randomized participants receiving at least one dose of correct study medication. One participant received both 25 mg and 50 mg doses during the study and was excluded from all analyses.
Groups:
- Placebo: After an observation period of ~5 weeks, participants receive dose-matched placebo to odanacatib once weekly for 52 weeks. Participants also receive weekly supplementation with open-label 5600 IU vitamin D3 and 500 mg of open-label daily calcium supplement (if calcium <1000 mg per day from dietary and other sources) throughout the observation and treatment periods.
- Total: Total of all reporting groups
Arm/Group | Placebo | Odanacatib 10 mg | Odanacatib 25 mg | Odanacatib 50 mg | Total
Number analyzed (Participants) | 73 | 74 | 70 | 69 | 286
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.7 (6.8) | 69.1 (7.3) | 67.5 (7.4) | 68.7 (7.0) | 68.2 (7.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 70 | 69 | 63 | 67 | 269
  Male | 3 | 5 | 7 | 2 | 17

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline to Week 52 in Lumbar Spine Bone Mineral Density (BMD) at Lumbar Vertebrae 1 to 4 (L1-L4)
Description: BMD (g/cm2) data was measured by dual-energy X-ray absorptiometry (DXA) at lumbar spine vertebrae 1 through 4 (L1-L4) from anterior view at the Observation visit (up to 5 weeks before Treatment Period), Week 0 (start of Treatment Period) and Week 52 (end of Treatment Period) or at discontinuation. Baseline was defined as the average of the 2 values collected at the Observation visit and Week 0 visit. Percent change from baseline in BMD = ([BMD at Week 52 visit] - [baseline BMD] ÷ baseline BMD) × 100. Measurements were performed using the Hologic Quantitative Digital Radiography (QDR) Series densitometer, and by same machine and under same scan mode throughout the study period. BMD data was centrally judged.
Time Frame: Baseline (Observation visit to Wk 0 treatment visit), Week 52
Population: Full Analysis Set (FAS): All randomized participants receiving at least one dose of study medication and with necessary on-treatment lumbar spine BMD measurements, with data carried forward.
Measure: Least Squares Mean (95% Confidence Interval); unit: percent change
Arm/Group | Placebo | Odanacatib 10 mg | Odanacatib 25 mg | Odanacatib 50 mg
Number analyzed (Participants) | 69 | 73 | 70 | 68
percent change | 0.55 [-0.32 to 1.42] | 4.09 [3.24 to 4.93] | 5.67 [4.81 to 6.54] | 5.94 [5.07 to 6.82]
Statistical Analysis 1: Comparison: Placebo vs Odanacatib 50 mg; Analysis for percent change from baseline to Week 52 in BMD was performed using a stepwise linear contrast test based on an analysis of covariance (ANCOVA) model with terms for treatment and study center. Treatment effect was assessed by Least-Squares means (LS mean) and the associated 95% confidence intervals. Estimated difference from placebo = odanacatib dose minus placebo dose. Positive mean treatment differences were in favor of odanacatib; Test type: Superiority or Other; p < 0.001, ANCOVA — The stepwise linear trend test adjusted for multiplicity within the family of comparisons of active doses with placebo and preserved the Type I error rate. P-value is for Placebo through Odanacatib 50 mg dose; Difference in LS Means = 5.40, 95% CI 2-sided [4.16 to 6.64]
Statistical Analysis 2: Comparison: Placebo vs Odanacatib 25 mg; Analysis for percent change from baseline to Week 52 in BMD was performed using a stepwise linear contrast test based on an ANCOVA model with terms for treatment and study center. Treatment effect was assessed by LS mean and the associated 95% confidence intervals. Estimated difference from placebo = odanacatib dose minus placebo dose. Positive mean treatment differences were in favor of odanacatib; Test type: Superiority or Other; p < 0.001, ANCOVA — The stepwise linear trend test adjusted for multiplicity within the family of comparisons of active doses with placebo and preserved the Type I error rate. P-value is for Placebo through Odanacatib 25 mg dose; Difference in LS Means = 5.12, 95% CI 2-sided [3.90 to 6.35]
Statistical Analysis 3: Comparison: Placebo vs Odanacatib 10 mg; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p < 0.001, ANCOVA — The stepwise linear trend test adjusted for multiplicity within the family of comparisons of active doses with placebo and preserved the Type I error rate. P-value is for Placebo through Odanacatib 10 mg dose; Difference in LS Means = 3.54, 95% CI 2-sided [2.33 to 4.75]

2. Secondary Outcome: Percent Change From Baseline to Week 52 in Total Hip BMD
Description: BMD (g/cm2) data was measured by DXA for total hip at the Observation visit (up to 5 weeks before Treatment Period), Week 0 (start of Treatment Period) and Week 52 (end of Treatment Period) or at discontinuation. Baseline was defined as the average of the 2 values collected at the Observation visit and Week 0 visit. Percent change from baseline in BMD = ([BMD at Week 52 visit] - [baseline BMD] ÷ baseline BMD) × 100. Measurements were performed using the Hologic QDR Series densitometer, and by same machine and under same scan mode throughout the study period. BMD data was centrally judged.
Time Frame: Baseline (Observation visit to Wk 0 treatment visit), Week 52
Population: FAS: All randomized participants receiving at least one dose of study medication and with necessary on-treatment total hip BMD measurements, with data carried forward.
Measure: Least Squares Mean (95% Confidence Interval); unit: percent change
Arm/Group | Placebo | Odanacatib 10 mg | Odanacatib 25 mg | Odanacatib 50 mg
Number analyzed (Participants) | 71 | 74 | 70 | 68
percent change | -0.35 [-1.00 to 0.29] | 1.31 [0.68 to 1.94] | 1.85 [1.20 to 2.50] | 2.70 [2.05 to 3.36]
Statistical Analysis 1: Comparison: Placebo vs Odanacatib 50 mg; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Difference in LS Means = 3.06, 95% CI 2-sided [2.14 to 3.98]
Statistical Analysis 2: Comparison: Placebo vs Odanacatib 25 mg; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 1, analysis 2]; Difference in LS Means = 2.20, 95% CI 2-sided [1.29 to 3.12]
Statistical Analysis 3: Comparison: Placebo vs Odanacatib 10 mg; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 1, analysis 3]; Difference in LS Means = 1.67, 95% CI 2-sided [0.77 to 2.57]

3. Primary Outcome: Number of Participants That Experienced an Adverse Event (AE)
Description: An AE was defined as any unfavorable and unintended change in the structure (sign), function (symptoms), or chemistry of the body (laboratory data) temporally associated with the use of the SPONSOR's products (including placebo), whether or not considered related to the use of the product. Any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a preexisting condition which is temporally associated with the use of the SPONSOR's product was also an AE. The number of participants that experienced at least one AE was reported for each treatment arm.
Time Frame: From first dose up to Post-Study (up to 54 weeks)
Population: Safety Population: All randomized participants receiving at least one dose of correct study medication. One participant received both 25 mg and 50 mg doses and was excluded from all analyses.
Measure: Number; unit: participants
Arm/Group | Placebo | Odanacatib 10 mg | Odanacatib 25 mg | Odanacatib 50 mg
Number analyzed (Participants) | 73 | 74 | 70 | 69
participants | 57 | 63 | 62 | 58

4. Primary Outcome: Number of Participants That Discontinued Study Drug Due to an AE
Description: An AE was defined as any unfavorable and unintended change in the structure (sign), function (symptoms), or chemistry of the body (laboratory data) temporally associated with the use of the SPONSOR's products (including placebo), whether or not considered related to the use of the product. Any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a preexisting condition which is temporally associated with the use of the SPONSOR's product was also an AE. The number of participants that discontinued study drug due to an AE was reported for each treatment arm. Participants may have discontinued study drug but continued on the trial.
Time Frame: From first dose up to end of treatment (up to 52 weeks)
Population: as for outcome 3
Measure: Number; unit: participants
Arm/Group | Placebo | Odanacatib 10 mg | Odanacatib 25 mg | Odanacatib 50 mg
Number analyzed (Participants) | 73 | 74 | 70 | 69
participants | 3 | 2 | 1 | 1

5. Secondary Outcome: Percent Change From Baseline to Week 52 in Femoral Neck BMD
Description: BMD (g/cm2) data was measured by DXA at the femoral neck subregion of the hip at the Observation visit (up to 5 weeks before Treatment Period), Week 0 (start of Treatment Period) and Week 52 (end of Treatment Period) or at discontinuation. Baseline was defined as the average of the 2 values collected at the Observation visit and Week 0 visit. Percent change from baseline in BMD = ([BMD at Week 52 visit] - [baseline BMD] ÷ baseline BMD) × 100. Measurements were performed using the Hologic QDR Series densitometer, and by same machine and under same scan mode throughout the study period. BMD data was centrally judged.
Time Frame: Baseline (Observation visit to Wk 0 treatment visit), Week 52
Population: FAS: All randomized participants receiving at least one dose of study medication and with necessary on-treatment femoral neck BMD measurements, with data carried forward.
Measure: Least Squares Mean (95% Confidence Interval); unit: percent change
Arm/Group | Placebo | Odanacatib 10 mg | Odanacatib 25 mg | Odanacatib 50 mg
Number analyzed (Participants) | 71 | 74 | 70 | 68
percent change | -0.72 [-1.58 to 0.13] | 1.51 [0.67 to 2.35] | 1.14 [0.27 to 2.00] | 2.35 [1.47 to 3.23]
Statistical Analysis 1: Comparison: Placebo vs Odanacatib 50 mg; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Difference in LS Means = 3.08, 95% CI 2-sided [1.85 to 4.31]
Statistical Analysis 2: Comparison: Placebo vs Odanacatib 25 mg; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.003, ANCOVA — [p-value comment as in outcome 1, analysis 2]; Difference in LS Means = 1.86, 95% CI 2-sided [0.64 to 3.08]
Statistical Analysis 3: Comparison: Placebo vs Odanacatib 10 mg; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 1, analysis 3]; Difference in LS Means = 2.23, 95% CI 2-sided [1.03 to 3.43]

6. Secondary Outcome: Percent Change From Baseline to Week 52 in Trochanter BMD
Description: BMD (g/cm2) data was measured by DXA at the trochanter subregion of the hip (near bony protrusions along outside edge of femur) at the Observation visit (up to 5 weeks before Treatment Period), Week 0 (start of Treatment Period) and Week 52 (end of Treatment Period) or at discontinuation. Baseline was defined as the average of the 2 values collected at the Observation visit and Week 0 visit. Percent change from baseline in BMD = ([BMD at Week 52 visit] - [baseline BMD] ÷ baseline BMD) × 100. Measurements were performed using the Hologic QDR Series densitometer, and by same machine and under same scan mode throughout the study period. BMD data was centrally judged.
Time Frame: Baseline (Observation visit to Wk 0 treatment visit), Week 52
Population: FAS: All randomized participants receiving at least one dose of study medication and with necessary on-treatment trochanter BMD measurements, with data carried forward.
Measure: Least Squares Mean (95% Confidence Interval); unit: percent change
Arm/Group | Placebo | Odanacatib 10 mg | Odanacatib 25 mg | Odanacatib 50 mg
Number analyzed (Participants) | 71 | 74 | 70 | 68
percent change | -0.28 [-1.31 to 0.76] | 2.16 [1.14 to 3.17] | 3.56 [2.52 to 4.60] | 4.38 [3.33 to 5.44]
Statistical Analysis 1: Comparison: Placebo vs Odanacatib 50 mg; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Difference in LS Means = 4.66, 95% CI 2-sided [3.18 to 6.14]
Statistical Analysis 2: Comparison: Placebo vs Odanacatib 25 mg; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 1, analysis 2]; Difference in LS Means = 3.84, 95% CI 2-sided [2.37 to 5.30]
Statistical Analysis 3: Comparison: Placebo vs Odanacatib 10 mg; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.002, ANCOVA — [p-value comment as in outcome 1, analysis 3]; Difference in LS Means = 2.43, 95% CI 2-sided [0.99 to 3.88]

7. Secondary Outcome: Percent Change From Baseline to Week 52 in Urinary N-telopeptides/Creatinine (u-NTx/Cre) Ratio
Description: The u-NTx/Cre ratio is a biochemical marker index of bone resorption. Urine samples were collected from second void morning urine specimens to assess the u-NTx/Cre ratio. Percent change from baseline in biomarker = ([biomarker value at Week 52 visit] - [baseline biomarker value] ÷ baseline biomarker value) × 100. All measurements of bone biochemical markers were centrally performed.
Time Frame: Baseline (Wk 0), Week 52
Population: Per Protocol (PP) Population: All randomized participants receiving at least one dose of study medication, who complied with the protocol (excludes participants with major protocol violation), and with available u-NTx/Cre data.
Measure: Least Squares Mean (95% Confidence Interval); unit: percent change
Arm/Group | Placebo | Odanacatib 10 mg | Odanacatib 25 mg | Odanacatib 50 mg
Number analyzed (Participants) | 50 | 57 | 56 | 51
percent change | -7.84 [-21.19 to 7.76] | -43.59 [-51.26 to -34.71] | -52.16 [-58.73 to -44.54] | -58.48 [-64.42 to -51.54]
Statistical Analysis 1: Comparison: Placebo vs Odanacatib 50 mg; The log-transformed fraction from baseline in biomarker levels was analyzed using an ANCOVA model with terms for treatment and study center, using a stepwise linear contrast test based on the ANCOVA model. The geometric mean percent change from baseline (back-transformation from the mean log-transformed fraction) and the associated 95% confidence intervals were presented; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Difference in LS Means = -50.64, 95% CI 2-sided [-66.43 to -34.84]
Statistical Analysis 2: Comparison: Placebo vs Odanacatib 25 mg; [analysis description as in outcome 7, analysis 1]; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 1, analysis 2]; Difference in LS Means = -44.32, 95% CI 2-sided [-60.42 to -28.21]
Statistical Analysis 3: Comparison: Placebo vs Odanacatib 10 mg; [analysis description as in outcome 7, analysis 1]; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 1, analysis 3]; Difference in LS Means = -35.75, 95% CI 2-sided [-52.33 to -19.16]

8. Secondary Outcome: Percent Change From Baseline to Week 52 in Serum C-Telopeptides of Type 1 Collagen (s-CTx) Level
Description: s-CTx is a biochemical marker index of bone resorption. Blood samples were collected in the morning and in fasting state for measurement of s-CTx. Percent change from baseline in biomarker = ([biomarker value at Week 52 visit] - [baseline biomarker value] ÷ baseline biomarker value) × 100. All measurements of bone biochemical markers were centrally performed.
Time Frame: Baseline (Wk 0), Week 52
Population: PP Population: All randomized participants receiving at least one dose of study medication, who complied with the protocol (excludes participants with major protocol violation), and with available s-CTx data.
Measure: Least Squares Mean (95% Confidence Interval); unit: percent change
Arm/Group | Placebo | Odanacatib 10 mg | Odanacatib 25 mg | Odanacatib 50 mg
Number analyzed (Participants) | 50 | 57 | 56 | 52
percent change | -10.95 [-32.05 to 16.72] | -49.68 [-60.92 to -35.20] | -71.64 [-78.04 to -63.39] | -71.36 [-78.02 to -62.68]
Statistical Analysis 1: Comparison: Placebo vs Odanacatib 50 mg; [analysis description as in outcome 7, analysis 1]; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Difference in LS Means = -60.42, 95% CI 2-sided [-85.70 to -35.13]
Statistical Analysis 2: Comparison: Placebo vs Odanacatib 25 mg; [analysis description as in outcome 7, analysis 1]; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 1, analysis 2]; Difference in LS Means = -60.70, 95% CI 2-sided [-85.91 to -35.49]
Statistical Analysis 3: Comparison: Placebo vs Odanacatib 10 mg; [analysis description as in outcome 7, analysis 1]; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 1, analysis 3]; Difference in LS Means = -38.73, 95% CI 2-sided [-65.94 to -11.52]

9. Secondary Outcome: Percent Change From Baseline to Week 52 in Urinary Deoxypyridinoline/Creatinine Ratio (u-DPD/Cre)
Description: The u-DPD/Cre ratio is a biochemical marker index of bone resorption. Urine samples were collected from second void morning urine specimens to assess the u-DPD/Cre ratio. Percent change from baseline in biomarker = ([biomarker value at Week 52 visit] - [baseline biomarker value] ÷ baseline biomarker value) × 100. All measurements of bone biochemical markers were centrally performed.
Time Frame: Baseline (Wk 0), Week 52
Population: PP Population: All randomized participants receiving at least one dose of study medication, who complied with the protocol (excludes participants with major protocol violation), and with available u-DPD/Cre data.
Measure: Least Squares Mean (95% Confidence Interval); unit: percent change
Arm/Group | Placebo | Odanacatib 10 mg | Odanacatib 25 mg | Odanacatib 50 mg
Number analyzed (Participants) | 50 | 57 | 56 | 51
percent change | 16.45 [-1.24 to 37.30] | -10.32 [-23.11 to 4.61] | -21.00 [-32.39 to -7.69] | -26.46 [-37.51 to -13.46]
Statistical Analysis 1: Comparison: Placebo vs Odanacatib 50 mg; [analysis description as in outcome 7, analysis 1]; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Difference in LS Means = -42.91, 95% CI 2-sided [-65.55 to -20.27]
Statistical Analysis 2: Comparison: Placebo vs Odanacatib 25 mg; [analysis description as in outcome 7, analysis 1]; Test type: Superiority or Other; p = 0.001, ANCOVA — [p-value comment as in outcome 1, analysis 2]; Difference in LS Means = -37.45, 95% CI 2-sided [-60.32 to -14.59]
Statistical Analysis 3: Comparison: Placebo vs Odanacatib 10 mg; [analysis description as in outcome 7, analysis 1]; Test type: Superiority or Other; p = 0.017, ANCOVA — [p-value comment as in outcome 1, analysis 3]; Difference in LS Means = -26.77, 95% CI 2-sided [-50.37 to -3.16]

10. Secondary Outcome: Percent Change From Baseline to Week 52 in Serum Bone Specific Alkaline Phosphatase (s-BSAP) Level
Description: s-BSAP is a biochemical marker index of bone formation. Blood samples were collected in the morning and in fasting state for measurement of s-BSAP. Percent change from baseline in biomarker = ([biomarker value at Week 52 visit] - [baseline biomarker value] ÷ baseline biomarker value) × 100. All measurements of bone biochemical markers were centrally performed.
Time Frame: Baseline (Wk 0), Week 52
Population: PP Population: All randomized participants receiving at least one dose of study medication, who complied with the protocol (excludes participants with major protocol violation), and with available s-BSAP data.
Measure: Least Squares Mean (95% Confidence Interval); unit: percent change
Arm/Group | Placebo | Odanacatib 10 mg | Odanacatib 25 mg | Odanacatib 50 mg
Number analyzed (Participants) | 53 | 60 | 58 | 54
percent change | -9.91 [-17.02 to -2.20] | -7.44 [-14.31 to -0.02] | -22.47 [-28.32 to -16.14] | -25.43 [-31.26 to -19.12]
Statistical Analysis 1: Comparison: Placebo vs Odanacatib 50 mg; [analysis description as in outcome 7, analysis 1]; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Difference in LS Means = -15.52, 95% CI 2-sided [-25.11 to -5.93]
Statistical Analysis 2: Comparison: Placebo vs Odanacatib 25 mg; [analysis description as in outcome 7, analysis 1]; Test type: Superiority or Other; p = 0.009, ANCOVA — [p-value comment as in outcome 1, analysis 2]; Difference in LS Means = -12.55, 95% CI 2-sided [-22.16 to -2.94]
Statistical Analysis 3: Comparison: Placebo vs Odanacatib 10 mg; [analysis description as in outcome 7, analysis 1]; Test type: Superiority or Other; p = 0.598, ANCOVA — [p-value comment as in outcome 1, analysis 3]; Difference in LS Means = 2.48, 95% CI 2-sided [-7.79 to 12.74]

11. Secondary Outcome: Percent Change From Baseline to Week 52 in Serum N-Terminal Propeptides of Type 1 Collagen (s-P1NP) Level
Description: s-P1NP is a biochemical marker index of bone formation. Blood samples were collected in the morning and in fasting state for measurement of s- P1NP. Percent change from baseline in biomarker = ([biomarker value at Week 52 visit] - [baseline biomarker value] ÷ baseline biomarker value) × 100. All measurements of bone biochemical markers were centrally performed.
Time Frame: Baseline (Wk 0), Week 52
Population: PP Population: All randomized participants receiving at least one dose of study medication, who complied with the protocol (excludes participants with major protocol violation), and with available s-P1NP data.
Measure: Least Squares Mean (95% Confidence Interval); unit: percent change
Arm/Group | Placebo | Odanacatib 10 mg | Odanacatib 25 mg | Odanacatib 50 mg
Number analyzed (Participants) | 53 | 60 | 58 | 54
percent change | -20.14 [-32.74 to -5.18] | -25.75 [-36.81 to -12.76] | -48.99 [-56.71 to -39.90] | -47.00 [-55.28 to -37.19]
Statistical Analysis 1: Comparison: Placebo vs Odanacatib 50 mg; [analysis description as in outcome 7, analysis 1]; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Difference in LS Means = -26.86, 95% CI 2-sided [-43.30 to -10.42]
Statistical Analysis 2: Comparison: Placebo vs Odanacatib 25 mg; [analysis description as in outcome 7, analysis 1]; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 1, analysis 2]; Difference in LS Means = -28.86, 95% CI 2-sided [-44.97 to -12.75]
Statistical Analysis 3: Comparison: Placebo vs Odanacatib 10 mg; [analysis description as in outcome 7, analysis 1]; Test type: Superiority or Other; p = 0.458, ANCOVA — [p-value comment as in outcome 1, analysis 3]; Difference in LS Means = -5.61, 95% CI 2-sided [-23.79 to 12.56]

ADVERSE EVENTS:
Time Frame: From first dose up to Post-Study (up to 54 weeks)
Description: Safety Population: All randomized participants receiving at least one dose of correct study medication. One participant received both 25 mg and 50 mg doses and was excluded from all analyses.
Arm/Group | Placebo | Odanacatib 10 mg | Odanacatib 25 mg | Odanacatib 50 mg
Serious Adverse Events (participants affected / at risk) | 5/73 | 6/74 | 4/70 | 4/69
Other Adverse Events (participants affected / at risk) | 46/73 | 46/74 | 50/70 | 51/69
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=73) | Odanacatib 10 mg (N=74) | Odanacatib 25 mg (N=70) | Odanacatib 50 mg (N=69)
Angina pectoris (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Myocardial ischaemia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Cataract (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ileus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Radius fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Foot deformity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cerebellar haemorrhage (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Intraneural cyst (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Subarachnoid haemorrhage (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neurosis (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=73) | Odanacatib 10 mg (N=74) | Odanacatib 25 mg (N=70) | Odanacatib 50 mg (N=69)
Abdominal discomfort (Gastrointestinal disorders) | 2 (3) | 0 (0) | 1 (2) | 4 (5)
Constipation (Gastrointestinal disorders) | 4 (4) | 4 (5) | 8 (9) | 6 (6)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 2 (2) | 3 (3) | 5 (6)
Gastritis (Gastrointestinal disorders) | 2 (2) | 4 (5) | 1 (1) | 1 (1)
Periodontitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 4 (4) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 5 (6) | 3 (3) | 2 (2) | 0 (0)
Bronchitis (Infections and infestations) | 4 (4) | 1 (1) | 2 (3) | 2 (2)
Cystitis (Infections and infestations) | 3 (3) | 1 (1) | 5 (5) | 7 (11)
Gastroenteritis (Infections and infestations) | 4 (4) | 0 (0) | 2 (2) | 0 (0)
Nasopharyngitis (Infections and infestations) | 22 (33) | 25 (36) | 26 (36) | 25 (39)
Pharyngitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 5 (7)
Contusion (Injury, poisoning and procedural complications) | 2 (2) | 4 (4) | 4 (4) | 2 (4)
Joint sprain (Injury, poisoning and procedural complications) | 5 (5) | 2 (2) | 2 (3) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 4 (4)
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 (5) | 0 (0) | 5 (7) | 3 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 7 (8) | 8 (8) | 10 (11) | 5 (5)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 4 (5) | 6 (6) | 10 (11) | 5 (5)
Periarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 2 (2) | 5 (6)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 4 (4) | 3 (4) | 4 (4) | 2 (3)
Dizziness (Nervous system disorders) | 5 (9) | 2 (2) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 3 (4) | 5 (5) | 1 (1) | 1 (1)
Eczema (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1) | 4 (4) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 4 (10) | 0 (0) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The SPONSOR must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication/presentation. Any information identified by the SPONSOR as confidential must be deleted prior to submission. SPONSOR review can be expedited to meet publication guidelines.